CLINICAL TRIAL: NCT02367274
Title: Use Of A Point-Of-Care TBI Detection System For Identification Of Head Injured Patients Who Present To The Emergency Department
Brief Title: Point-Of-Care TBI Detection System For Head Injured Patients In The Emergency Department
Acronym: READ-TBI
Status: Completed | Type: Observational
Sponsor: BrainScope Company, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 11-Ahead
Record Dates: First submitted 2015-02-11; First posted 2015-02-20 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2015-12

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: BrainScope Ahead 200 — A single-use, proprietary headset containing pre-gelled electrodes will be placed on the subject's forehead according to the standard locations of the modified International 10/20 system. Subjects will undergo approximately 5 minutes of eyes closed brain electrical activity recording.

SUMMARY:
A prospective, non-randomized trial for the extension and replication of the development database of brain electrical activity recordings and clinical information collected from patients who present to the ED following closed head injury.

DETAILED DESCRIPTION:
The objective of this study is to test the clinical utility of the BrainScope technology for the acute identification of traumatic structural brain injury in the TBI population, following closed head injury. The data generated will serve to validate and/or refine the current algorithms to detect acute, traumatic, structural brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are admitted to the ED and are suspected of a traumatic, closed head injury within 24 hours. The patient will have a GCS 12-15 upon arrival to the ED even if GCS was lower prior to arrival to the ED (e.g., at the time of injury).

Exclusion Criteria:

* Subjects will be excluded who have forehead, scalp, or skull abnormalities or other conditions that would prevent correct application of the electrode headset on the skin.
* In addition,

  * subjects with dementia,
  * Parkinson's Disease,
  * multiple sclerosis,
  * seizure disorder,
  * brain tumors,
  * history of brain surgery,
  * psychiatric disorder being managed by a psychiatric healthcare professional/provider,
  * substance dependence,
  * history of TIA or stroke within the last year,
  * currently receiving dialysis or in end-stage renal disease,
  * active fever defined as greater than 100 degrees F or 37.7 degrees C,
  * current condition is "critical" in the opinion of the investigator,
  * subject is suffering from an open head injury,
  * subject requires advanced airway management (i.e. mechanical ventilation), currently receiving procedural sedation medications.
* Subjects below the age of 18 years, and prisoners will not be eligible for study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are suspected of a traumatic, closed head injury within 24 hours will be recruited from patients who enter the Emergency Department at hospitals that are participating as clinical sites for this study.
Sampling Method: Non-Probability Sample
Enrollment: 421 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Extend and replicate a database of brain electrical activity and clinical information collected from patients who present to the ED following closed head injury | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Douglas C Oberly, Principal Investigator — BrainScope Company, Inc.
Locations (11):
- United States (11):
  - Hartford Hospital, Hartford, Connecticut
  - Emory University- Grady Hospital, Atlanta, Georgia
  - R Cowley Shock Trauma Hospital, Baltimore, Maryland
  - Wayne State University - Detroit Receiving Hospital, Detroit, Michigan
  - Wayne State University - Sinai Grace Hospital, Detroit, Michigan
  - Washington University - Barnes Jewish Hospital, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - UT-Houston Health Science Center, Houston, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia

REFERENCES:
- [Background] Huff JS, Jahar S. Differences in interpretation of cranial computed tomography in ED traumatic brain injury patients by expert neuroradiologists. Am J Emerg Med. 2014 Jun;32(6):606-8. doi: 10.1016/j.ajem.2014.03.010. Epub 2014 Mar 18. PMID 24731934
- [Background] Prichep LS, Naunheim R, Bazarian J, Mould WA, Hanley D. Identification of hematomas in mild traumatic brain injury using an index of quantitative brain electrical activity. J Neurotrauma. 2015 Jan 1;32(1):17-22. doi: 10.1089/neu.2014.3365. PMID 25054838
- [Background] O'Neil B, Naunheim R, DeLorenzo R. CT positive brain injury in mild TBI patients presenting with normal SAC scores. Mil Med. 2014 Nov;179(11):1250-3. doi: 10.7205/MILMED-D-13-00585. PMID 25373049
- [Background] Prichep LS, Jacquin A, Filipenko J, Dastidar SG, Zabele S, Vodencarevic A, Rothman NS. Classification of traumatic brain injury severity using informed data reduction in a series of binary classifier algorithms. IEEE Trans Neural Syst Rehabil Eng. 2012 Nov;20(6):806-22. doi: 10.1109/TNSRE.2012.2206609. Epub 2012 Jul 26. PMID 22855231
- [Background] Prichep LS, Ghosh Dastidar S, Jacquin A, Koppes W, Miller J, Radman T, O'Neil B, Naunheim R, Huff JS. Classification algorithms for the identification of structural injury in TBI using brain electrical activity. Comput Biol Med. 2014 Oct;53:125-33. doi: 10.1016/j.compbiomed.2014.07.011. Epub 2014 Aug 1. PMID 25137412
- [Result] Naunheim RS, Treaster M, English J, Casner T. Automated electroencephalogram identifies abnormalities in the ED. Am J Emerg Med. 2011 Oct;29(8):845-8. doi: 10.1016/j.ajem.2010.03.010. Epub 2010 May 1. PMID 20825903
- [Result] O'Neil B, Prichep LS, Naunheim R, Chabot R. Quantitative brain electrical activity in the initial screening of mild traumatic brain injuries. West J Emerg Med. 2012 Nov;13(5):394-400. doi: 10.5811/westjem.2011.12.6815. PMID 23359586
- [Result] Naunheim RS, Treaster M, English J, Casner T, Chabot R. Use of brain electrical activity to quantify traumatic brain injury in the emergency department. Brain Inj. 2010;24(11):1324-9. doi: 10.3109/02699052.2010.506862. PMID 20722504
- [Result] Hanley DF, Chabot R, Mould WA, Morgan T, Naunheim R, Sheth KN, Chiang W, Prichep LS. Use of brain electrical activity for the identification of hematomas in mild traumatic brain injury. J Neurotrauma. 2013 Dec 15;30(24):2051-6. doi: 10.1089/neu.2013.3062. Epub 2013 Nov 23. PMID 24040943
- [Result] Ayaz SI, Thomas C, Kulek A, Tolomello R, Mika V, Robinson D, Medado P, Pearson C, Prichep LS, O'Neil BJ. Comparison of quantitative EEG to current clinical decision rules for head CT use in acute mild traumatic brain injury in the ED. Am J Emerg Med. 2015 Apr;33(4):493-6. doi: 10.1016/j.ajem.2014.11.015. Epub 2014 Nov 20. PMID 25727167